CLINICAL TRIAL: NCT07359560
Title: Intravenous Lidocaine Versus Magnesium Sulfate for Hemodynamic Stability During Emergence From General Anesthesia in Infertility-related Laparoscopic Gynecologic Surgeries
Brief Title: Lidocaine vs Magnesium Sulfate for Hemodynamic Stability During Emergence in Infertility-Related Laparoscopic Surgery"
Acronym: LidoMagGyna
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amira S kenawy ,md, Lecturer of Anesthesia, Intensive Care, and Pain Management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZU-IRB# 1904/2-Nov -2025; ethics commitee approval numbe (Other: zagazig university faculty of medicine)
Record Dates: First submitted 2025-12-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Infertility Female; Hemodynamic Instability
Keywords: lidocaine magnisium; hemodynamic instability; infertility female; laparoscopic surgery
MeSH Terms: conditions — Infertility, Female | interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride; Saline Solution; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into three parallel groups to receive one of the study interventions (intravenous lidocaine, intravenous magnesium sulfate, or normal saline control). Each participant will receive only one intervention, and outcomes will be assessed independently for each group. Randomization and identical preparation of study drugs will maintain blinding of participants, anesthesia providers, and outcome assessors throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug preparations (lidocaine, magnesium sulfate, and normal saline) will be prepared in identical syringes and infusion bags by an anesthesiologist who is not involved in patient care or data collection. This ensures that participants, anesthesia care providers, investigators, and outcome assessors remain blinded to group allocation throughout the study. Randomization codes will be securely stored and will not be revealed until after data analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Control Group (Normal Saline) (Placebo Comparator): Participants in this arm will receive 15 mL of 0.9% normal saline intravenously over 15 minutes, starting 30 minutes before the anticipated time of extubation. This serves as the control intervention for comparison with lidocaine and magnesium sulfate.
  Interventions: Drug: Normal Saline (Intravenous)
- Arm 2: Lidocaine Group (Experimental): Participants in this arm will receive intravenous lidocaine at a dose of 1.5 mg/kg diluted with 0.9% normal saline to a total volume of 15 mL. The infusion will be administered over 15 minutes, starting 30 minutes before the expected time of extubation.
  Interventions: Drug: Lidocaine (drug)
- Arm 3: Magnesium Sulfate Group (Experimental): Participants in this arm will receive intravenous magnesium sulfate at a dose of 30 mg/kg diluted with 0.9% normal saline to a total volume of 15 mL. The infusion will be administered over 15 minutes, starting 30 minutes before the anticipated time of extubation.
  Interventions: Drug: magnesium sulfate

INTERVENTIONS:
Drug: Lidocaine (drug) — The intervention described in this clinical study involves a comparative prospective randomized double-blind controlled trial to assess the effects of intravenous Lidocaine versus Magnesium Sulfate compared to a Control group for hemodynamic stability during emergence from general anesthesia in infertility-related laparoscopic gynecologic surgeries.
  Other Names: magnisium sulfate; saline
  Arms: Arm 2: Lidocaine Group
Drug: Normal Saline (Intravenous) — 0.9% normal saline, total volume 15 mL, administered intravenously over 15 minutes starting 30 minutes before the anticipated time of extubation.
  Arms: Arm 1: Control Group (Normal Saline)
Drug: Lidocaine (drug) — Lidocaine 1.5 mg/kg diluted with 0.9% normal saline to a total volume of 15 mL, administered intravenously over 15 minutes starting 30 minutes before the anticipated time of extubation.
  Arms: Arm 2: Lidocaine Group
Drug: magnesium sulfate — Magnesium sulfate 30 mg/kg diluted with 0.9% normal saline to a total volume of 15 mL, administered intravenously over 15 minutes starting 30 minutes before the anticipated time of extubation.
  Arms: Arm 3: Magnesium Sulfate Group

SUMMARY:
This study is being conducted to compare two medications, intravenous lidocaine and intravenous magnesium sulfate, and their ability to keep blood pressure and heart rate stable during the period of waking up from general anesthesia in infertility-related laparoscopic gynecologic surgeries.

Laparoscopic gynecologic procedures can cause changes in heart rate and blood pressure, especially during emergence from anesthesia, and these changes may affect patient safety.

In this randomized, double-blind clinical trial, women scheduled for elective infertility-related laparoscopic surgery will be assigned to one of three groups: lidocaine, magnesium sulfate, or a control group. The study will evaluate mean arterial pressure (primary outcome), heart rate, pain scores, sedation level, nausea and vomiting, and any side effects during and after surgery.

The goal is to determine which medication provides better hemodynamic stability and improves recovery in the early postoperative period.

DETAILED DESCRIPTION:
Laparoscopic gynecologic procedures performed for infertility are commonly associated with significant changes in heart rate and blood pressure, especially during the emergence phase of general anesthesia. These hemodynamic fluctuations may increase the risk of discomfort, delayed recovery, or cardiovascular complications. Several medications, including lidocaine and magnesium sulfate, have been suggested to help stabilize these responses because of their analgesic, sympatholytic, and cardioprotective properties. However, there is limited evidence comparing the two drugs in this specific surgical population.This prospective, randomized, double-blind controlled trial aims to evaluate the effects of intravenous lidocaine and intravenous magnesium sulfate on hemodynamic stability during emergence from general anesthesia in women undergoing elective infertility-related laparoscopic gynecologic surgeries. Participants will be randomly assigned to one of three groups: a lidocaine group, a magnesium sulfate group, or a control group receiving normal saline. Study medications will be administered 30 minutes before the anticipated time of extubation.

Hemodynamic measurements will be recorded throughout the perioperative period, with particular focus on mean arterial pressure during emergence (primary outcome). Secondary measures include heart rate, postoperative pain scores, sedation levels, nausea and vomiting, and any adverse events observed within the first 24 hours after surgery. All patients will receive standardized anesthesia management, monitoring, and postoperative care.

The goal of the study is to identify which medication is more effective in maintaining stable hemodynamics and improving early recovery following laparoscopic gynecologic surgery for infertility.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 21 to 40 years

Body mass index (BMI) between 18.5 and 29 kg/m²

American Society of Anesthesiologists (ASA) physical status I or II

Scheduled for elective infertility-related laparoscopic gynecologic surgery (e.g., diagnostic laparoscopy, ovarian cystectomy, adhesiolysis) under general anesthesia

Expected duration of anesthesia less than 2 hours

Ability to provide written informed consent

Exclusion Criteria:

Known allergy or contraindication to lidocaine or magnesium sulfate

History of significant cardiac, renal, or hepatic disease

Chronic use of analgesics or history of drug dependence

History of myasthenia gravis

Pregnancy or positive serum β-hCG test

-

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The full title of the study is "Intravenous Lidocaine Versus Magnesium Sulfate for Hemodynamic Stability During Emergence From General Anesthesia in Infertility-Related Laparoscopic Gynecologic surgeries" , and the inclusion criteria focus on conditions and procedures unique to women
Enrollment: 69 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
the mean arterial pressure | 6 months
  MAP mean arterial pressure Measurement Schedule During Emergence MAP will be continuously monitored during the emergence phase of anesthesia. Recordings will be documented at minute 0 (the exact moment of extubation) and 5 minutes after extubation, starting from 5 minutes before extubation

SECONDARY OUTCOMES:
heart rate | Preoperative: Baseline HR measurement. Intraoperative: 5 minutes after intubation. After Trendelenburg position. After pneumoperitoneum. Every 5 minutes for 30 minutes after infusion of lidocaine or magnesium sulfate. Emergence from Anesthesia:
  HR heart rate serves as an important measure to determine how well the interventions (lidocaine or magnesium sulfate) manage hemodynamic stability during the delicate phase of emergence from anesthesia.
Visual Analog Scale (VAS) for Pain | Visual Analog Scale (VAS) for Pain 30 minutes, 2 hours, and 6 hours postoperatively
  Pain intensity assessed using the Visual Analog Scale (VAS), a 10-cm scale ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater pain intensity.
Ramsay Sedation Score | Preoperative (if applicable): Baseline sedation status. Postoperative (PACU): On arrival in PACU: To assess the initial recovery from anesthesia. 30 minutes after arrival in PACU: To evaluate recovery progress and sedation changes. 6 hours postoperat
  assess the sedation level in patients recovering from general anesthesia during the postoperative period.The Ramsey Sedation Score is a 6-point scale used to assess the depth of sedation in patients. The score is based on the patient's responsiveness to verbal commands and physical stimuli, which allows clinicians to monitor sedation levels effectively.
Incidence of Hypotension: | Immediately after induction of anesthesia (post-intubation): Blood pressure (MAP) will be measured to ensure the patient's cardiovascular system is stable after anesthesia induction. After placement in Trendelenburg position (head-down position): Th
  A decrease in Mean Arterial Pressure (MAP) by more than 20% from the baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Kenawy, lecturer, Principal Investigator — Zagazig University Hospitals, Zagazig University
Locations (1):
- Zagazig University Faculty of Medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is single-center, data contain sensitive patient information, and participant-level access is not planned."